CLINICAL TRIAL: NCT04018872
Title: A Phase II Trial Evaluating the Effectiveness of Itraconazole in Improving Pathologic Complete Response Rates in Patients With Esophageal Cancer Through Inhibition of the Hedgehog and AKT Signaling Pathways
Brief Title: Evaluating the Effect of Itraconazole on Pathologic Complete Response Rates in Esophageal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dallas VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, David Wang, Staff Physician, Dallas VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-017
Record Dates: First submitted 2019-07-10; First posted 2019-07-15 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Esophagus Adenocarcinoma; Esophagus Squamous Cell Carcinoma; Gastroesophageal Junction Adenocarcinoma
Keywords: itraconazole; esophageal neoplasms; esophagus; esophagogastric junction; adenocarcinoma; squamous cell carcinoma
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms; Adenocarcinoma; Carcinoma, Squamous Cell | interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Itraconazole (Experimental): Itraconazole capsule 300mg twice daily for 6-8 weeks following chemoradation.
  Interventions: Drug: Itraconazole

INTERVENTIONS:
Drug: Itraconazole — Oral administration of itraconazole twice daily from completion of neoadjuvant chemoradiation until esophagectomy.

SUMMARY:
Esophageal cancer, which has a low 5-year overall survival rate for all stages (<20%) , is increasing in incidence. Previous studies have shown that the Hedgehog (Hh) and AKT signaling pathways are activated in a significant proportion of esophageal cancers. Itraconazole, a widely used anti-fungal medication, has been shown to inhibit various pathways involved in esophageal cancer tumorigenesis including Hh and AKT. In this phase II clinical trial, the investigators aim to evaluate the effect of itraconazole as a neoadjuvant therapy following standard of care chemoradiation in the treatment of locoregional esophageal and gastroesophageal junction carcinomas.

DETAILED DESCRIPTION:
Esophageal cancer has a high incidence rate in the United States, and novel approaches to its treatment are being studied. Itraconazole, an antifungal agent, has been shown to inhibit the Hedgehog (Hh) and AKT signaling pathways, which are upregulated in esophageal cancer and promote tumor cell growth. This study will evaluate whether the use of itraconazole leads to increased rates of pathological complete response (pathCR) by at least 15% from the historical pathCR rate of 25% in patients with esophageal cancer or gastroesophageal junction (GEJ) adenocarcinoma. The investigators will enroll approximately 78 patients with esophageal cancer or GEJ adenocarcinoma who will then undergo standard of care staging work-up with a PET/CT and endoscopic ultrasound (EUS). In a subset of patients, biopsies will be obtained to assess the status of the Hh and AKT signaling pathways by PCR, Western blot, and immunohistochemistry in the primary tumor before treatment. If no distant metastases are found, all patients will undergo 5-6 weeks of standard of care neoadjuvant chemoradiation. Following this, all patients will be given itraconazole 300 mg twice daily for 6-8 weeks. Adverse effects to itraconazole will be monitored in oncology clinic. If standard restaging PET/CT following neoadjuvant chemoradiation does not reveal new metastases, the patient will undergo an esophagectomy. Samples from normal esophageal tissue will be analyzed for presence of itraconazole and its metabolites to determine if the patients were taking the study drug. Tumor tissue will be evaluated for status of Hh pathway activation, AKT and VEGFR2 phosphorylation, Ki67 immunostaining, and other molecular pathways with comparisons made to pre-treatment biopsies if available. The final pathology report will indicate whether the patient has achieved pathCR. Because the Hh signaling pathway is a resistance pathway that can be upregulated in response to chemoradiation, the investigators believe that administering itraconazole following neoadjuvant chemoradiation will lead to a higher pathCR rate. This in turn should be able to improve treatment outcomes in patients with esophageal cancer and GEJ adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with localized (locoregional) esophageal cancer
* Patients diagnosed with localized (locoregional) gastroesophageal junction cancer

Exclusion Criteria:

* Patients unwilling or unable to provide informed consent
* Patients with QTc>450ms
* Patients with a history of symptomatic congestive heart failure
* Patients with LFT's>3xULN
* Patients who are pregnant
* Patients with a known allergy to itraconazole

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2019-06-24 (Actual); Primary Completion 2026-06-24 (Estimated); Study Completion 2026-09-29 (Estimated)

PRIMARY OUTCOMES:
Percentage of pathological complete response with itraconazole | 3-4 months
  Generally for esophageal cancer the pathological complete response rate at time of esophagectomy is 25%, and we have designed our study with the projected number of patients assuming we observe an improvement of 15% or more in this rate following treatment with itraconazole. This is the study's primary endpoint. By inhibiting the Hh signaling pathway with the use of itraconazole, we anticipate improved pathological complete response rates.

SECONDARY OUTCOMES:
Comparison of hedgehog biomarkers before and after intervention | 3-4 months
  As part of clinical staging, patients will undergo endoscopic ultrasound (EUS) following a PET/CT that does not show metastases. During EUS, some patients will undergo eight research biopsies obtained with large forceps for research purposes at the level of the visualized esophageal mass or abnormality (3 for RNA isolation, 3 for protein isolation, and 2 for formalin fixation). Three research biopsies for RNA isolation will also be obtained from normal appearing esophagus, at least 5 cm away from any mass lesions. The research biopsies will be submitted to qPCR analysis for mRNA expression levels of SHH, IHH, PTCH, GLI1, GLI2, and GLI3 (Hedgehog pathway components). Comparisons will be made between mass biopsies and normal esophageal tissues. Following esophagectomy, tissues will be analyzed for the aforementioned hedgehog pathway markers to determine response to therapy.
Comparison of phosphorylated VEGFR2 and AKT before and after intervention | 3-4 months
  Tissue obtained prior to initiation of chemoradiation will be analyzed with Western blot to quantify presence of VEGFR2 and AKT. These markers will again be analyzed following esophagectomy to determine response to therapy.
Levels of itraconazole and metabolites in esophageal tissue | 1 month.
  The concentration of itraconazole and hydroxy-itraconazole in normal esophageal tissue will be measured following esophagectomy to ensure that the drug has been taken consistently.

CONTACTS AND LOCATIONS:
Overall Officials: David Wang, MD, PhD, Principal Investigator — North Texas Veterans Healthcare System
Locations (1):
- Dallas VA Medical Center, Dallas, Texas, United States

REFERENCES:
- [Background] Kim DJ, Kim J, Spaunhurst K, Montoya J, Khodosh R, Chandra K, Fu T, Gilliam A, Molgo M, Beachy PA, Tang JY. Open-label, exploratory phase II trial of oral itraconazole for the treatment of basal cell carcinoma. J Clin Oncol. 2014 Mar 10;32(8):745-51. doi: 10.1200/JCO.2013.49.9525. Epub 2014 Feb 3. PMID 24493717
- [Background] Antonarakis ES, Heath EI, Smith DC, Rathkopf D, Blackford AL, Danila DC, King S, Frost A, Ajiboye AS, Zhao M, Mendonca J, Kachhap SK, Rudek MA, Carducci MA. Repurposing itraconazole as a treatment for advanced prostate cancer: a noncomparative randomized phase II trial in men with metastatic castration-resistant prostate cancer. Oncologist. 2013;18(2):163-73. doi: 10.1634/theoncologist.2012-314. Epub 2013 Jan 22. PMID 23340005
- [Background] Nacev BA, Grassi P, Dell A, Haslam SM, Liu JO. The antifungal drug itraconazole inhibits vascular endothelial growth factor receptor 2 (VEGFR2) glycosylation, trafficking, and signaling in endothelial cells. J Biol Chem. 2011 Dec 23;286(51):44045-44056. doi: 10.1074/jbc.M111.278754. Epub 2011 Oct 24. PMID 22025615
- [Background] Kim J, Tang JY, Gong R, Kim J, Lee JJ, Clemons KV, Chong CR, Chang KS, Fereshteh M, Gardner D, Reya T, Liu JO, Epstein EH, Stevens DA, Beachy PA. Itraconazole, a commonly used antifungal that inhibits Hedgehog pathway activity and cancer growth. Cancer Cell. 2010 Apr 13;17(4):388-99. doi: 10.1016/j.ccr.2010.02.027. PMID 20385363
- [Background] Chen MB, Liu YY, Xing ZY, Zhang ZQ, Jiang Q, Lu PH, Cao C. Itraconazole-Induced Inhibition on Human Esophageal Cancer Cell Growth Requires AMPK Activation. Mol Cancer Ther. 2018 Jun;17(6):1229-1239. doi: 10.1158/1535-7163.MCT-17-1094. Epub 2018 Mar 28. PMID 29592879